CLINICAL TRIAL: NCT00931840
Title: A Phase 2 Study of EZN-2208 (PEG-SN38) Administered With or Without Cetuximab in Patients With Metastatic Colorectal Carcinoma (mCRC)
Brief Title: A Study of EZN-2208 Administered With or Without Cetuximab in Patients With Metastatic Colorectal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EZN-2208-04
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: EZN-2208 (PEG-SN38)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — EZN-2208; Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EZN-2208 (Experimental): EZN-2208 will be administered as an i.v. infusion on weekly basis for 3 weeks and repeated every 28 days.
  PLEASE NOTE THAT ENROLLMENT IN EXPERIMENTAL ARM (ARM A) IS COMPLETE. NO NEW PATIENT IN THIS ARM IS ALLOWED TO ENROLL.
  Interventions: Drug: EZN-2208, Cetuximab and Irinotecan
- Cetuximab + EZN-2208 (Experimental): Cetuximab will be administered as an i.v. infusion on weekly basis. EZN-2208 administered as i.v. infusion on weekly basis for 3 weeks and repeated every 28 days.
  Interventions: Drug: EZN-2208, Cetuximab and Irinotecan
- Irinotecan + cetuximab (Active Comparator): Cetuximab will be administered weekly as an i.v. infusion. Irinotecan will be administered as an i.v. infusion on Weeks 1 and 2 and repeated every 3 weeks.
  Interventions: Drug: EZN-2208, Cetuximab and Irinotecan

INTERVENTIONS:
Drug: EZN-2208, Cetuximab and Irinotecan — Patients with mutated K RAS tumors will be treated with single-agent EZN-2208 (Arm A). PLEASE NOTE THAT ENROLLMENT IN EXPERIMENTAL ARM (ARM A) IS COMPLETE. NO NEW PATIENT IN THIS ARM IS ALLOWED TO ENROLL.
  Patients with wild-type K-RAS tumors will be randomly assigned in a 2:1 ratio to EZN-2208 + cetuximab (Arm B) or the benchmark of irinotecan + cetuximab (Arm C).
  Other Names: Irinotecan, (CPT 11),(Camptosar®); Erbitux (cetuximab)

SUMMARY:
This is a Phase 2, multicenter, multiple-arm, open-label study to evaluate the efficacy, safety, and tolerability of EZN-2208. EZN-2208 will be administered as a single agent in patients with K-RAS mutations in the tumors. Patients with wild type K-RAS in tumors will be randomized to EZN-2208 + cetuximab or to standard of care (Camptosar® + cetuximab), patients must have failed regimens containing irinotecan (Camptosar®, CPT-11), oxaliplatin (Eloxatin®), and fluoropyrimidine.

After discontinuation of study treatment, patients will receive care as considered appropriate by the investigator. Patients will continue to be followed for disease progression, subsequent anticancer therapy, and survival.

DETAILED DESCRIPTION:
EZN-2208 will be administered by i.v. infusion weekly for 3 weeks in 4-week cycles. The cetuximab infusion will be administered before the EZN-2208 (Arm B) or irinotecan (Arm C) infusion. Study treatment will be continued until evidence of disease progression, unacceptable toxicity, or withdrawal of the patient's consent for participation in the study.

Approximately 220 patients will be enrolled in this study: approximately 100 patients in the K-RAS mutated arm and approximately 120 patients in the wild-type K-RAS arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be eligible for enrollment in the study.

  1. Histologically confirmed CRC adenocarcinoma that is metastatic or locally recurrent CRC that is nonresectable
  2. Patients must agree to genetic testing of the original or metastatic CRC tumor biopsy tissue for K-RAS mutational status.
  3. Disease progression
  4. Previous therapy with irinotecan, oxaliplatin, and fluoropyrimidine either alone or in any combination(s). Patients must have radiographically documented progressive disease while receiving, or within 3 months of receiving, these agents alone or in combination.
  5. No more than 2 prior cytotoxic chemotherapy regimens.
  6. Age 18 years or older
  7. Measurable disease by RECIST Version 1.1
  8. ECOG performance status of 0 or 1
  9. Adequate bone marrow, renal, and hepatic function

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria will not be eligible for enrollment.

  1. Known chronic infectious disease
  2. Major surgery within 3 weeks before study start
  3. Known or suspected brain metastases requiring intervention with steroids and/or radiation therapy.
  4. Prior chemotherapy, immunotherapy, non-investigational agent, or other therapy used to treat the cancer within 3 weeks before the scheduled administration of EZN-2208
  5. History of other primary cancer within 5 years of enrollment, unless

     1. Curatively resected non-melanomatous skin cancer, or
     2. Curatively resected cervical cancer
  6. Lack of recovery to Grade 1 from any reversible side effects related to the administration of an investigational agent, or other prior treatments for the cancer
  7. Any condition such as uncontrollable diabetes, uncontrollable hypertension, or active infection.
  8. Current participation in another clinical study with an investigational agent and/or use of an investigational drug (not including investigational use of an approved drug) in the 30 days before the first administration of EZN-2208

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-10 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 2011

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 2011

CONTACTS AND LOCATIONS:
Overall Officials: Richard M. Goldberg, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (60):
- United States (35):
  - Location #033, Tucson, Arizona
  - Location# 042, Alhambra, California
  - Location # 043, Bakersfield, California
  - Location# 044, Fullerton, California
  - Location# 019, La Jolla, California
  - Location# 046, Long Beach, California
  - Location# 053, Los Angeles, California
  - Location# 051, Northridge, California
  - Location# 045, Pomona, California
  - Location # 048, Santa Barbara, California
  - Location # 049, Santa Barbara, California
  - Location# 052, Santa Maria, California
  - Location #027, Stanford, California
  - Location# 003, Newark, Delaware
  - Location# 047, Orlando, Florida
  - Location# 022, Port Saint Lucie, Florida
  - Location# 005, Marietta, Georgia
  - Location# 009, Chicago, Illinois
  - Location #050, Terre Haute, Indiana
  - Location# 029, Worcester, Massachusetts
  - Location #031, Lebanon, New Hampshire
  - Location # 030, Buffalo, New York
  - Location# 035, New York, New York
  - Location# 002, New York, New York
  - Location# 007, The Bronx, New York
  - Location# 001, Chapel Hill, North Carolina
  - Location# 020, Goldsboro, North Carolina
  - Location# 024, Winston-Salem, North Carolina
  - Location# 008, Columbus, Ohio
  - Location# 037, Lancaster, Pennsylvania
  - Location# 018, Greenville, South Carolina
  - Location# 004, Memphis, Tennessee
  - Location #038, Houston, Texas
  - Location# 011, Lubbock, Texas
  - Location# 021, San Antonio, Texas
- Canada (5):
  - Location# 076, Ottawa, Ontario
  - Location # 079, Toronto, Ontario
  - Location# 077, Montreal, Quebec
  - Location# 074, Montreal, Quebec
  - Location# 055, Rimouski, Quebec
- Israel (8):
  - Location# 066, Tel-Aviv, Central District
  - Location# 071, Kfar Saba, Sharon
  - Location# 072, Beersheba, South District
  - Location# 068, Be’er Ya‘aqov
  - Location# 067, Haifa
  - Location# 073, Jerusalem District
  - Location# 070, Tel Aviv
  - Location# 069, Tel Litwinsky
- Netherlands (2):
  - Location# 041, Leiden, NL
  - Location # 040, Rotterdam, The Netherlands
- United Kingdom (10):
  - Location #065, Dorchester, Dorset
  - Location # 083, London, England
  - Location# 057, London, Greater London
  - Location# 054-2, London, Greater London
  - Location #061, London, Greater London
  - Location# 064, Manchester, Greater Manchester
  - Location# 056, Edinburgh, Scotland
  - Location# 062, Glasgow, Scotland
  - Location# 054, Sutton, Surrey
  - Location# 063, Leeds, West Yorkshire